CLINICAL TRIAL: NCT01135602
Title: Topiramate for Hospitalized Patients With Alcoholism: a 12-Week Open-Label Study
Brief Title: Topiramate for Hospitalized Patients With Alcoholism: a 12-week Study
Acronym: THoPA-O
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Manit Srisurapanont, Department of Psychiatry, Faculty of Medicine, Chiang Mai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THoPA-O
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2010-06

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcoholism; Topiramate
MeSH Terms: conditions — Alcoholism | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topiramate (Experimental): 1 group
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Topiramate 50-300 mg/day Orally Twice per day
  Other Names: Topamax

SUMMARY:
12-week, open-label study of topiramate in hospitalized patients with alcoholism

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized due to alcohol-related problems
* DSM-IV-TR alcohol dependence
* >/= 35 drinks/week (male) or >/= 28 drinks/week (female) for >/= 1 week during four weeks prior to the admission
* AUDIT score >/= 8
* Mild or no alcohol withdrawal
* Body mass index > 18 kg/m2
* No pregnancy and no plan for pregnancy (female)
* Intention to decrease or stop drinking

Exclusion Criteria:

* Severe psychiatric and cognitive disorders
* Other substance dependence, except nicotine and caffeine dependence, during 6 months prior to enrollment
* Taking antipsychotics, mood stabilizers, anticonvulsants, opioid analgesics, systematic steroids, carbonic anhydrase inhibitors, hydrochlorthiazide, metformin, pioglitazone, or disulfiram
* Moderate to high risk of suicide
* Medical history of narrow angle glaucoma, renal impairment, kidney stones, and seizures
* Unstable medical conditions
* Plan to receive a formal treatment for alcoholism from other treatment settings
* Under legal process
* Pregnancy and nursing woman
* Abnormal laboratory tests, including blood urea nitrogen, creatinine, electrolytes, and fasting blood sugar

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Cognition | 12 weeks
  Cognition will be assessed by the use of Montreal Cognitive Assessment (MoCA)

SECONDARY OUTCOMES:
Alcohol drink/day | 12 weeks
  Alcohol drink/day assessed by the use of Timeline Followback (TLFB)

CONTACTS AND LOCATIONS:
Overall Officials: Manit Srisurapanont, MD, Principal Investigator — Department of Psychiatry, Faculty of Medicine, Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai, Thailand